CLINICAL TRIAL: NCT01403168
Title: Comparative Evaluation of Osteopathy Treatment Efficacy in Pain Support After Breast Surgery in Oncology
Acronym: OSTEOPATHIE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSTEOPATHIE
Record Dates: First submitted 2011-07-21; First posted 2011-07-27 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: Osteopathy; Breast cancer; Pain
MeSH Terms: conditions — Breast Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- osteopathy + conventional analgesic treatments (Experimental)
  Interventions: Other: OSTEOPATHY + conventional analgesic treatments
- conventional analgesic treatments (Placebo Comparator)
  Interventions: Other: Conventional analgesic treatments

INTERVENTIONS:
Other: OSTEOPATHY + conventional analgesic treatments — 5 sessions for osteopathy are planned and will start in the 15 days following the enrollment.
  The conventional analgesic treatments will be administered in the 15 days following the enrollment.
  Arms: osteopathy + conventional analgesic treatments
Other: Conventional analgesic treatments — These treatments will be administered in the 15 days following the enrollment. Dose and frequence will depend on patients.
  Arms: conventional analgesic treatments

SUMMARY:
This is an open, prospective, controlled, randomized, comparative study with 2 arms.

The purpose of the study is to assess the efficacy of osteopathy after breast surgery.

80 patients will be enrolled, 40 per arm. Patients will be randomized at inclusion and will be followed during one year.

ELIGIBILITY:
Inclusion Criteria:

* woman >= 18 years
* pain (median VAS >=3 on the week prior to inclusion)
* mastectomy or tumorectomy with axillary dissection <= 12 months
* PS <=2
* able to write, understand and read French
* signed informed consent

Exclusion Criteria:

* no pain
* immediate breast reconstruction
* history of cognitive or psychiatric troubles

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-04; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of the osteopathy treatment on pain | 3 months
  Pain is assessed by means of visual analogic scale (from 0 to 10 points). A decrease of 2 points after 3 months is expected.

CONTACTS AND LOCATIONS:
Overall Officials: Gisele CHVETZOFF, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France

REFERENCES:
- [Background] Fassoulaki A, Patris K, Sarantopoulos C, Hogan Q. The analgesic effect of gabapentin and mexiletine after breast surgery for cancer. Anesth Analg. 2002 Oct;95(4):985-91, table of contents. doi: 10.1097/00000539-200210000-00036. PMID 12351281
- [Background] Ivens D, Hoe AL, Podd TJ, Hamilton CR, Taylor I, Royle GT. Assessment of morbidity from complete axillary dissection. Br J Cancer. 1992 Jul;66(1):136-8. doi: 10.1038/bjc.1992.230. PMID 1637663
- [Background] Jung BF, Ahrendt GM, Oaklander AL, Dworkin RH. Neuropathic pain following breast cancer surgery: proposed classification and research update. Pain. 2003 Jul;104(1-2):1-13. doi: 10.1016/s0304-3959(03)00241-0. No abstract available. PMID 12855309
- [Background] Labreze L, Dixmerias-Iskandar F, Monnin D, Bussieres E, Delahaye E, Bernard D, Lakdja F. [Postmastectomy pain syndrome evidence based guidelines and decision trees]. Bull Cancer. 2007 Mar;94(3):275-85. French. PMID 17371770
- [Background] Dirks J, Fredensborg BB, Christensen D, Fomsgaard JS, Flyger H, Dahl JB. A randomized study of the effects of single-dose gabapentin versus placebo on postoperative pain and morphine consumption after mastectomy. Anesthesiology. 2002 Sep;97(3):560-4. doi: 10.1097/00000542-200209000-00007. PMID 12218520
- [Background] Eija K, Tiina T, J NP. Amitriptyline effectively relieves neuropathic pain following treatment of breast cancer. Pain. 1996 Feb;64(2):293-302. doi: 10.1016/0304-3959(95)00138-7. PMID 8740607
- [Background] Attal N, Cruccu G, Haanpaa M, Hansson P, Jensen TS, Nurmikko T, Sampaio C, Sindrup S, Wiffen P; EFNS Task Force. EFNS guidelines on pharmacological treatment of neuropathic pain. Eur J Neurol. 2006 Nov;13(11):1153-69. doi: 10.1111/j.1468-1331.2006.01511.x. PMID 17038030
- [Background] Vick DA, McKay C, Zengerle CR. The safety of manipulative treatment: review of the literature from 1925 to 1993. J Am Osteopath Assoc. 1996 Feb;96(2):113-5. doi: 10.7556/jaoa.1996.96.2.113. PMID 8838907
- [Background] Ernst E. Manipulation of the cervical spine: a systematic review of case reports of serious adverse events, 1995-2001. Med J Aust. 2002 Apr 15;176(8):376-80. doi: 10.5694/j.1326-5377.2002.tb04459.x. PMID 12041633
- [Background] Licht PB, Christensen HW, Hoilund-Carlsen PF. Is cervical spinal manipulation dangerous? J Manipulative Physiol Ther. 2003 Jan;26(1):48-52. doi: 10.1067/mmt.2003.42. PMID 12532139
- [Background] Vickers A, Zollman C. ABC of complementary medicine. The manipulative therapies: osteopathy and chiropractic. BMJ. 1999 Oct 30;319(7218):1176-9. doi: 10.1136/bmj.319.7218.1176. No abstract available. PMID 10541511
- [Background] Noll DR, Degenhardt BF, Stuart M, McGovern R, Matteson M. Effectiveness of a sham protocol and adverse effects in a clinical trial of osteopathic manipulative treatment in nursing home patients. J Am Osteopath Assoc. 2004 Mar;104(3):107-13. No abstract available. PMID 15083985
- [Background] Hayes NM, Bezilla TA. Incidence of iatrogenesis associated with osteopathic manipulative treatment of pediatric patients. J Am Osteopath Assoc. 2006 Oct;106(10):605-8. PMID 17122030